CLINICAL TRIAL: NCT03373396
Title: Impact of Chlordecone Exposure on Evolution of Fibrosis to Cirrhosis in Chronic Hepatitis C, B or Alcoholic, in Guadeloupe.
Brief Title: Impact of Chlordecone on Active Chronic Hepatitis
Acronym: HEPATOCHLORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBM-PAP-2011/25
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Fibrosis, Liver
Keywords: Chlordecone; fibrosis; cirrhosis; chronic hepatitis B, C; alcohol; viral hepatitis; transaminases; fibroscan
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Hepatitis B, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: It is a case-control study. There will be two groups. The patient will be assigned to a group according to the Metavir classification. F0 patients will be in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group with Metavir score between F1 and F4 (Other): Patient with Metavir score between F1 and F4 will be assigned to the case group. Collected data will contain epidemiological and biological data, blood samples with chlordecone dosage.
  Interventions: Diagnostic Test: Blood samples
- Control group with Metavir score of between F0 (Other): Patient with Metavir score of F0 will be assigned to the control group. Collected data will contain epidemiological and biological data. Blood samples with chlordecone dosage will be performed.
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — Collected data will contain epidemiological and biological data, blood samples with chlordecone dosage.

SUMMARY:
Chlordecone is known to induce liver damage in rat and mice but no data exists in human being. However chlordecone was used until 1993 in French West Indies for banana fields, it is important to test what damage can be induced now, for patients exposed. We should consider chlordecone as a potential cofactor of liver fibrosis. So we have chosen to compare two populations of chronic hepatitis B, C or alcoholic, with cirrhosis or without fibrosis due to active hepatitis, who had been exposed to chlordecone.

DETAILED DESCRIPTION:
Actually, there is no data concerning the impact of chlordecone on the evolution of fibrosis to cirrhosis in chronic hepatitis whereas many studies have been reported liver damage in mice. The goal of this study is to know if co-exposition to chlordecone can induce evolution to cirrhosis in chronic hepatitis due to alcohol or viral hepatitis. At first, we will assess a group of patients with chronic hepatitis B, C or due to alcohol without fibrosis. And they will be compared to patients with cirrhosis exposed to chlordecone too. Patients will be included in 2 hospital centers. All these patients should have an active liver disease. The activity will be defined by histology or elevated transaminases (>2N), fibrosis will be defined by histology or an association of fibroscan and biological markers. Exposition to chlordecone will be evaluated by a blood chlordecone measure for every patient.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Active chronic hepatitis B or C or alcoholic
* Patient without previous antiviral therapy, activity confirmed by histology or elevated transaminases
* Alcohol consumption more than 20g/d for women and 30g/d for men responsible of chronic alcoholic disease
* Seronegative HIV status, inform consent signed, health insurance

Exclusion Criteria:

* Inactive chronic hepatitis
* Other chronic hepatitis as auto-immune hepatitis, hemochromatosis, wilson disease, acute hepatitis due to medication, transplantation, antiviral or imunosupressive treatment, psychiatric disease
* Co-infection with HIV, HBV or HCV
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2011-11-08 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2015-12-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of progression to cirrhosis with a correlation test between chlordecone exposure and fibrosis in active and chronic hepatitis due to virus B, C or alcohol. | through study completion, an average of 5 years.
  : Chlordecone level will be compared among the two groups (patients with or without significant fibrosis) in order to determine the impact of chlordecone on the evolution of fibrosis. Patients of each group will be paired according to the age, sex, origin of the liver disease. Analysis will be performed using SPSS software.

SECONDARY OUTCOMES:
Epidemiological study of hepatitis B, C and alcoholic in Guadeloupe | through study completion, an average of 5 years.
  Distribution of the main etiologies of chronic hepatitis according to age, sex and origin and severity of the liver disease for patients of each group will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Moana GELU SIMEON, hepato-gastoenterology, Principal Investigator — Hospital University Center of Pointe-à-Pitre
Locations (1):
- Hospital University Center of Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gelu-Simeon M, Lafrance MJ, Michineau L, Saillard E, Thome JP, Emond C, Samson M, Multigner L. Inverse association between plasma chlordecone concentrations and progression of alcoholic liver fibrosis: the role of liver metabolism. Environ Health. 2024 Mar 20;23(1):30. doi: 10.1186/s12940-024-01054-6. PMID 38504260